CLINICAL TRIAL: NCT06337838
Title: Bleeding Reduction in Acute and Chronic KidnEy patienTs Having Surgery (BRACKETS) Pilot Trial
Acronym: BRACKETS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024.BRACKETS-Pilot
Record Dates: First submitted 2024-01-22; First posted 2024-03-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Acute Kidney Injury; Bleeding; Surgery
Keywords: Major Noncardiac Surgery; Tranexamic Acid; Desmopressin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Hemorrhage | interventions — Deamino Arginine Vasopressin; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: 2x2 partial factorial design where patients are first randomized to receive prophylactic intravenous TXA versus placebo, and (when the study drug is available) to be randomized to receive prophylactic intravenous desmopressin versus placebo before noncardiac surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drugs will be sourced locally and will be prepared by appropriately qualified center personnel who are independent of the study team to ensure blinding is maintained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prophylactic intravenous tranexamic acid and prophylactic intravenous desmopressin. (Experimental): Within 20 minutes preceding anticipated skin incision, patients will receive preoperative prophylactic intravenous tranexamic acid at a dose of 1000 mg infused over 10 minutes for patients with estimated glomerular filtration rate (eGFR) <25 ml/min/1.73m2 who do not receive dialysis before surgery and 500 mg infused over 10 minutes for patients who receive dialysis.
  Within 20 minutes preceding anticipated skin incision, patients allocated to the desmopressin intervention group will receive intravenous desmopressin at a dose of 20 mcg over 30 minutes.
  Interventions: Drug: Desmopressin Injectable Solution; Drug: Tranexamic Acid Injectable Product
- Prophylactic intravenous tranexamic acid and placebo. (Experimental): Within 20 minutes preceding anticipated skin incision, patients will receive preoperative prophylactic intravenous tranexamic acid at a dose of 1000 mg infused over 10 minutes for patients with eGFR <25 ml/min/1.73m2 who do not receive dialysis before surgery and 500 mg infused over 10 minutes for patients who receive dialysis.
  Within 20 minutes preceding anticipated skin incision, patients allocated to the desmopressin control group will receive an intravenous infusion of 0.9% saline solution, administered over a duration of 30 minutes.
  Interventions: Drug: Tranexamic Acid Injectable Product; Other: Placebo
- Prophylactic intravenous desmopressin and placebo. (Experimental): Within 20 minutes preceding anticipated skin incision, patients will receive intravenous desmopressin at a dose of 20 mcg over 30 minutes. Patients will not receive prophylactic tranexamic acid.
  Within 20 minutes preceding anticipated skin incision, patients allocated to the tranexamic acid control group will receive an intravenous infusion of 0.9% saline solution. This saline solution will be administered over a duration of 10 minutes in a volume equivalent to that received by patients in the tranexamic acid intervention group.
  Interventions: Drug: Desmopressin Injectable Solution; Other: Placebo
- Placebo and placebo. (Placebo Comparator): Within 20 minutes preceding anticipated skin incision, patients allocated to the tranexamic acid control group will receive an intravenous infusion of 0.9% saline solution. This saline solution will be administered over a duration of 10 minutes in a volume equivalent to that received by patients in the tranexamic acid intervention group.
  Within 20 minutes preceding anticipated skin incision, patients allocated to the desmopressin control group will receive an intravenous infusion of 0.9% saline solution, administered over a duration of 30 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Desmopressin Injectable Solution — Intravenous desmopressin, 20 mcg, single dose administration.
  Other Names: DDAVP
  Arms: Prophylactic intravenous desmopressin and placebo.; Prophylactic intravenous tranexamic acid and prophylactic intravenous desmopressin.
Drug: Tranexamic Acid Injectable Product — Intravenous tranexamic acid, 1000 mg single dose administration for patients with eGFR<25 not yet receiving dialysis OR 500 mg single dose administration for patients receiving dialysis.
  Other Names: Cyklokapron
  Arms: Prophylactic intravenous tranexamic acid and placebo.; Prophylactic intravenous tranexamic acid and prophylactic intravenous desmopressin.
Other: Placebo — Intravenous 0.9% saline solution
  Arms: Placebo and placebo.; Prophylactic intravenous desmopressin and placebo.; Prophylactic intravenous tranexamic acid and placebo.

SUMMARY:
The BRACKETS pilot study is a multicentre, prospective, randomized controlled trial of prophylactic preoperative tranexamic acid (TXA) versus placebo and, using a partial factorial design, of prophylactic preoperative desmopressin versus placebo.

DETAILED DESCRIPTION:
Perioperative administration of TXA reduces bleeding risk in surgical patients. However, large clinical trials have excluded patients with advanced kidney disease, so the benefits remain uncertain in this population, and there is potential for harm. The benefit of desmopressin, which is purported to more directly address the defect of primary hemostasis believed important in severe kidney disease more directly than TXA, has not been examined in adequate randomized control trials (RCTs). Both medications are generic and have been available for many years. To convincingly test these medications in patients with severe kidney disease, large, global trials are required. This pilot-phase trial will 1) inform the feasibility and design of a large international trial to evaluate the efficacy and safety of TXA and desmopressin in patients with advanced kidney disease undergoing noncardiac surgery, 2) provide preliminary data regarding the efficacy and safety of TXA and desmopressin in people with advanced kidney disease having noncardiac surgery, and 3) provide pharmacokinetic data to inform dose selection.

ELIGIBILITY:
Eligibility criteria specific to the tranexamic acid (TXA) factorial component of trial Inclusion Criteria:

1. One of either:

   1.1. eGFR <25 ml/min/1.73m2 estimated using the CKD-Epi 2009 or 2021creatinine-based equation from the most recent serum creatinine measurement done in the previous 6 months; or 1.2. Receipt of dialysis (including hemodialysis, peritoneal dialysis, hemofiltration, or hemodiafiltration) within the last 7 days;
2. Planned noncardiac surgery (elective, urgent, or emergency surgery);
3. Expected to require at least an overnight hospital admission after surgery;
4. Age ≥18 years; and
5. Informed consent is obtained to participate in the BRACKETS-Pilot Trial.

Exclusion Criteria:

1. Undergoing cardiac surgery;
2. Undergoing intracranial neurosurgery;
3. Undergoing surgery for creation or revision of arteriovenous fistula or graft for dialysis access;
4. Planned use of prophylactic systemic TXA or ϵ-aminocaproic acid;
5. Hypersensitivity or known allergy to TXA;
6. History of seizure disorder;
7. Recent (within 90 days) stroke, myocardial infarction, acute arterial thrombosis, deep venous thrombosis, pulmonary embolism, or thrombosis of an arteriovenous fistula or graft;
8. History of thrombotic thrombocytopenic purpura, atypical hemolytic uremic syndrome, or antiphospholipid antibody syndrome;
9. Women who are known to be pregnant, breastfeeding, or who meet both of the following criteria: i) are of childbearing potential and do not have a negative pregnancy test documented in the 7 days before surgery, AND ii) are not using effective contraception; or
10. Previously enrolled in the BRACKETS-Pilot Trial.

Eligibility criteria specific to the desmopressin factorial component of trial

Inclusion criteria:

1. Included in the TXA factorial.

Exclusion criteria:

1. The hospital does not have access to desmopressin;
2. Planned use of prophylactic desmopressin;
3. Most recent serum sodium concentration < 130 mEq/L;
4. Known or suspected von Willebrand disease (any kind), hemophilia, or platelet function disorder; or
5. Hypersensitivity or known allergy to desmopressin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | Through study completion, an average of 1.5 years
  A rate of 0.25 patients per study site per week
Receipt of the allocated study drug within 1 hour before start of surgery for the tranexamic acid factorial | Day of surgery
  Account of whether the patient began to receive study drug for the TXA factorial within an hour before skin incision. Target ≥80% of participants
Receipt of the allocated study drug within 1 hour before start of surgery for the desmopressin factorial | Day of surgery
  Account of whether the patient began to receive study drug for the desmopressin factorial within an hour before skin incision. Target ≥80% of participants
Completion of 30-day follow-up | 30 days after randomization
  Account of whether the patient or their next-of-kin could be contacted and completed the 30-day post-randomization assessment. Target ≥80% of participants

SECONDARY OUTCOMES:
Bleeding Independently Associated with Mortality after noncardiac Surgery (BIMS) | 30 days after randomization
  Number of patients who experience BIMS
Bleeding Score | 30 days after randomization
  10-category ordinal score. Minimum scores mean a better outcome. 0 denotes no bleeding or bleeding in which the nadir hemoglobin is ≥70 g/L, no red blood transfusion was given, no reoperation for reasons of bleeding occurred, and there was no death imminently or directly caused by bleeding.
  1. denotes bleeding and post-operative hemoglobin <70 g/L or 1 unit of blood (red blood cells or whole blood) transfused.
  2. denotes bleeding and 2 units transfused.
  3. denotes bleeding and 3 units transfused.
  4. denotes bleeding and 4 units transfused
  5. denotes bleeding and 5 units transfused.
  6. denotes bleeding and 6 units transfused.
  7. denotes bleeding and 7 units transfused.
  8. denotes bleeding and 8 or more units of blood transfused.
  9. denotes reoperation for reasons of bleeding.
  10. denotes death imminently or directly caused by bleeding.
Reoperation for reasons of bleeding | 30 days after randomization
  Number of patients who return to the operating room for surgical management of suspected documented bleeding
Blood (red blood cells or whole blood) transfused | 30 days after randomization
  Number of units of blood transfused.
Blood (red blood cells or whole blood) transfused | Up to and including postoperative day 3 after surgery
  Number of units of blood transfused.
Any blood transfusion (red blood cells or whole blood) | 30 days after randomization
  Number of units of blood transfused.
Any blood transfusion (red blood cells or whole blood) | Up to and including postoperative day 3
  Number of units of blood transfused.
Lowest measured hemoglobin concentration | 30 days after randomization
  The mean absolute difference for continuous outcomes using linear regression with treatment allocation
Most recent hemoglobin concentration | 30 days after randomization
  The mean absolute difference for continuous outcomes using linear regression with treatment allocation
Death | 30 days after randomization
  Number of patients who die of any cause
Major arterial and venous thrombosis | 30 days after randomization
  (i.e., composite of myocardial injury after noncardiac surgery [MINS], stroke, peripheral arterial thrombosis, dialysis vascular access thrombosis requiring anticoagulation or intervention, and symptomatic venous thromboembolism)
Myocardial Injury after Noncardiac Surgery (MINS) | 30 days after randomization
  Number of patients who experience MINS
Myocardial Injury after Noncardiac Surgery (MINS) that meets criteria for myocardial infarction | 30 days after randomization
  Number of patients who experience MINS that meets criteria for myocardial infarction (based on the Fourth Universal Definition of myocardial infarction)
MINS that is an isolated ischemic troponin elevation | 30 days after randomization
  Number of patients who experience MINS that is an isolated ischemic troponin elevation
Stroke | 30 days after randomization
  Number of patients experiencing a stroke
Non-hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a non-hemorrhagic stroke
Hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a hemorrhagic stroke
Peripheral arterial thrombosis | 30 days after randomization
  Number of patients who experience a peripheral arterial thrombosis
Thrombosis of arteriovenous fistula or graft | 30 days after randomization
  Number of patients who have thrombosis of arteriovenous fistula or graft
Symptomatic proximal venous thromboembolism | 30 days after randomization
  Number of patients who experience symptomatic proximal venous thromboembolism
Symptomatic pulmonary embolism | 30 days after randomization
  Number of patients who experience a symptomatic pulmonary embolism
Symptomatic proximal leg or arm deep venous thrombosis (DVT) | 30 days after randomization
  Number of patients who experience a symptomatic proximal leg or arm DVT
Non-fatal cardiac arrest | 30 days after randomization
  Number of patients who experience non-fatal cardiac arrest
Coronary revascularization procedure | 30 days after randomization
  Number of patients who undergo coronary revascularization procedure
Clinically important atrial fibrillation or flutter | 30 days after randomization
  Number of patients who experience clinically important atrial fibrillation or flutter
Acute heart failure or clinically important volume overload | 30 days after randomization
  Number of patients who experience acute heart failure or clinically important volume overload.
Acute kidney injury (for patients not receiving dialysis before surgery) | 30 days after randomization
  Number of patients who experience an acute kidney injury
New start of dialysis | 30 days after randomization
  Number of patients who require new start of dialysis
Seizure | 30 days after randomization
  Number of patients who experience a seizure
Clinically significant intraoperative hypotension | 30 days after randomization
  Number of patients who experience clinically significant intraoperative hypotension
Clinically significant postoperative hypotension | Up to and including the end of postoperative day 1
  Number of patients who experience clinically significant postoperative hypotension
Sepsis | 30 days after randomization
  Number of patients who experience sepsis
Duration of surgery | 30 days after randomization
  The time from skin incision to closure, in minutes.
Receipt of platelets | 30 days after randomization
  Any transfusion of this blood product
Receipt of fibrinogen | 30 days after randomization
  Any transfusion of this blood product
Receipt of fresh frozen plasma | 30 days after randomization
  Any transfusion of this blood product
Receipt of cryoprecipitate | 30 days after randomization
  Any transfusion of this blood product
Receipt of recombinant Factor VIIa | 30 days after randomization
  Number of patients receiving recombinant factor VIIa
Receipt of prothrombin complex concentrate | 30 days after randomization
  Number of patients who receive prothrombin complex concentrate
Prescribed erythropoiesis stimulating agent | 30 days after randomization
  Number of patients receiving a weekly dose of erythropoiesis stimulating agent on prescription active at 30 days
Severe hyponatremia | Up to and including the end of postoperative day 1
  Measured serum sodium concentration <125 meq/L
Duration of hospital stay after surgery | Day of surgery and ending the day of discharge
  Cumulative number of nights spent in an acute care hospital
Duration of critical care stay after surgery | Day of surgery and ending the day of discharge
  Cumulative number of nights spent in an intensive care unit
Delayed graft function after kidney transplantation | Within 7 days following kidney transplantation
  Receipt of dialysis
Persistent dialysis dependence | 30 days after randomization
  Participant continues to receive dialysis after surgery.
Incisional site pain severity | 30 days after randomization in the last 24 hours
  Rating of pain using the 10-point ordinal scale where 0 corresponds to no pain and 10 corresponds to the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Roshanov, MC,MSc,FRCPC, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No